CLINICAL TRIAL: NCT06783166
Title: Assessing the Clinical Outcomes of Dapagliflozin Versus Acetazolamide in Patients With Acute Heart Failure
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha Mansour, Lecturer of Clinical Pharmacy, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS.24.04.2757
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Acute Heart Failure
MeSH Terms: interventions — dapagliflozin; Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin 10mg (Experimental): Patients will receive once daily dapagliflozin 10 mg orally in addition to loop diuretic therapy and standard care for 3 days.
  Interventions: Drug: Dapagliflozin 10mg
- Acetazolamide 500mg (Active Comparator): Patients will receive once daily acetazolamide 500 mg orally in addition to loop diuretic therapy and standard care for 3 days.
  Interventions: Drug: Acetazolamide 500mg

INTERVENTIONS:
Drug: Dapagliflozin 10mg — Dapagliflozin 10 mg is a medication classified as a sodium-glucose cotransporter-2 (SGLT-2) inhibitor.
  Arms: Dapagliflozin 10mg
Drug: Acetazolamide 500mg — Acetazolamide 500 mg is a medication classified as a carbonic anhydrase inhibitor.
  Arms: Acetazolamide 500mg

SUMMARY:
This study investigates the comparative clinical outcomes of dapagliflozin, an SGLT-2 inhibitor, versus acetazolamide, a carbonic anhydrase inhibitor, in patients hospitalized with acute heart failure (AHF). The trial aims to assess the effectiveness of these drugs in improving natriuretic and diuretic responses and shortening hospital stays. Dapagliflozin and acetazolamide will be added to standard loop diuretic therapy, and their safety profiles will be evaluated to identify potential side effects. This research seeks to provide evidence for incorporating these drugs into AHF management, with the potential to improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older who are hospitalized for hypervolemic AHF, with evidence of congestion defined as either:

   * 2 of the following signs or symptoms: peripheral edema, ascites, jugular venous pressure > 10mmHg, orthopnea, paroxysmal nocturnal dyspnea, 5-pound weight gain, or signs of congestion on chest x-ray or lung ultrasound. OR
   * If pulmonary artery catheterization is available, a pulmonary capillary wedge pressure greater than 19 mmHg plus a systemic physical exam finding of hypervolemia from the list above.
2. Randomized within 24 hours of hospitalization for AHF.
3. Planned use of IV loop diuretic therapy during current hospitalization
4. Estimated glomerular filtration rate (eGFR) of at least 30 ml/min/1.73m2 by the MDRD equation.

Exclusion Criteria:

1. Unable to follow instructions.
2. Treated with any proximal tubular diuretics.
3. Systolic blood pressure of less than 90 mm Hg.
4. An estimated glomerular filtration rate (GFR) of less than 20 ml per 1.73 m2 of body-surface area.
5. Type 1 diabetes mellitus.
6. Dyspnea is primarily due to non-cardiac causes.
7. Cardiogenic shock.
8. Acute coronary syndrome within 30 days prior to randomization.
9. Planned or recent percutaneous or surgical coronary intervention within 30 days prior to randomization.
10. Signs of ketoacidosis and/or hyperosmolar hyperglycemic syndrome (pH>7.30 and glucose >15 mmol/L and HCO3>18 mmol/L).
11. Pregnant or nursing (lactating) women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in dyspnea VAS (Visual analogue scale) | From baseline to day 3
  Comparing the area under the curve (AUC) of change in VAS dyspnea score. To do so, individual changes in VAS score will be visualized as a curve where the x-axis shows study day baseline to day 3, and y-axis shows VAS score. Using this approach, AUC for each study day will be calculated, and added together, resulting in an overall VAS AUC score (mm × h) that can be compared across treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Noha Mansour, PhD, Principal Investigator — Department of Clinical Pharmacy & Pharmacy Practice, Faculty of Pharmacy, University of Mansoura; Moheb Magdy Mouris, MD, Principal Investigator — Department of Cardiology, Faculty of Medicine, University of Mansoura; Mohamed El- Husseiny Shams, Professor, Study Chair — Department of Clinical Pharmacy & Pharmacy Practice, Faculty of Pharmacy, University of Mansoura
Locations (1):
- Noha Mansour, Al Mansurah, Egypt